CLINICAL TRIAL: NCT04231318
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of a Single Injection Cross-Linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide (Cingal®) to Provide Symptomatic Relief of Osteoarthritis of the Knee
Brief Title: Study of Cingal® and Triamcinolone Hexacetonide for the Relief of Knee Osteoarthritis Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cingal 19-01
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — 3,6,9,16,19,22-hexaaza-6,19-bis(2-hydroxyethyl)tricyclo(22,2,2,2(11,14))triaconta-1,11,13,24,27,29-hexaene; triamcinolone hexacetonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cingal (Experimental): Single injection of Cingal: 4 milliliter (mL) dose of 88 mg (22 mg/mL) of cross-linked sodium hyaluronate with 18 mg (4.5 mg/mL) of triamcinolone hexacetonide (TH). Manufactured by Anika Therapeutics.
  Interventions: Drug: Cingal
- Triamcinolone Hexacetonide (TH) (Active Comparator): Single injection of Triamcinolone Hexacetonide (TH): 1 milliliter (mL) dose of 20 mg/ml TH. Manufactured by IntraPharm.
  Interventions: Drug: Triamcinolone Hexacetonide (TH)
- Placebo (Placebo Comparator): Single injection of Placebo: 4 milliliter (mL) dose of 0.9% saline. Manufactured by Anika Therapeutics.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cingal — Single intra-articular injection of Cingal into the knee.
  Other Names: HA + TH
  Arms: Cingal
Drug: Triamcinolone Hexacetonide (TH) — Single intra-articular injection of TH into the knee.
  Other Names: TH
  Arms: Triamcinolone Hexacetonide (TH)
Drug: Placebo — Single intra-articular injection Placebo (0.9% Saline) into the knee.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, parallel group, placebo controlled trial to compare the safety and effectiveness of a single injection of Cingal® to a single injection of Triamcinolone Hexacetonide (TH) to achieve pain relief and other symptoms of osteoarthritis of the knee.

DETAILED DESCRIPTION:
To determine the contribution of Triamcinolone Hexacetonide (TH) when combined with sodium hyaluronate for pain relief, both in terms of magnitude and duration, when used as single injection, as compared to a single injection of TH alone in subjects diagnosed with osteoarthritis of the knee.

A saline placebo is included within the trial to set the expectation of a return to Baseline pain for the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 40-75 years old.
2. Body Mass Index (BMI) ≤ 40 kg/m2.
3. Subject has Kellgren-Lawrence (K-L) severity grade II or III in the Index knee as determined by X-Ray. Contralateral knee: K-L severity grade 0, I or II.
4. Subject has had at least two signs and at least two symptoms of OA disease (based on the European League Against Rheumatism (EULAR) recommendations for diagnosing knee OA) in the Index knee for at least 6 months despite conservative treatment (weight reduction, physical therapy, pain medications, etc.). The EULAR signs and symptoms are as follows:

   * Signs: crepitus, restricted movement and bony enlargement
   * Symptoms: persistent knee pain, limited morning stiffness and reduced function
5. Subject must be willing to abstain from other IA treatments of the knee for the duration of the study.
6. Subject is willing to discontinue all analgesics including nonsteroidal anti-inflammatory drugs (NSAIDs), except acetaminophen before the treatment injection and through the completion of the study. NSAIDs should be discontinued through the Screening period.
7. Subject is willing to use only acetaminophen (up to a maximum of 3.0 grams per day) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up visit, the Subject is willing to discontinue use of acetaminophen
8. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing ICF.
9. Subject is able to understand and comply with the requirements of the study and voluntarily provides consent.

Baseline Inclusion Criteria 24 Subject has a Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain-sub-score ≥ 50 mm and ≤ 90 mm in the affected knee and ≤ 30 mm in the contralateral knee on a 100 mm Visual Analog Scale (VAS) scale.

Exclusion Criteria:

1. Subject received an IA injection of Hyaluronic Acid (HA) and/or steroid in either knee within 6 months of signing the ICF. A Subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either knee during the course of this study.
2. Subject had an arthroscopy of either knee within 3 months of signing the ICF.
3. Subject had an open surgical procedure of either knee or hip or any surgery of the spine within 12 months of signing ICF. Subject plans to have knee, hip or spine surgery within the study period.
4. Subject has intra-articular trauma to the Index knee. Subject has concurrent multi-system or multi-limb trauma.
5. Subject has evidence or medical history of the following diseases in the Index knee: septic arthritis; inflammatory joint disease; history of Reiter's syndrome; gout; chondrocalcinosis associated with recurrent episodes of acute synovitis of the knee consistent with pseudogout; osteochondritis dissecans, Paget disease of the bone; ochronosis; acromegaly; hemochromatosis; primary osteochondromatosis; known history of Wilson disease; heritable disorders or collagen gene mutations.
6. Subject has a history of cartilage repair surgery in the Index knee within 3 years of signing the ICF.
7. Subject has a history of Anterior cruciate ligament (ACL) repair, reconstruction or injury in the Index knee within 3 years of signing the ICF.
8. Subject has X-Ray findings of acute fractures, severe bone loss, avascular necrosis, severe bone or joint deformity in the Index knee.
9. Subject has significant varus or valgus deformity greater than 8 degrees in either knee.
10. Subject has a clinically apparent tense effusion of the Index knee.
11. Subject has knee instability in either knee per the Investigator's assessment.
12. Subject requires consistent use of an assistive device (e.g. wheelchair, walker, etc.) Occasional use of a cane is acceptable.
13. Subject has medical condition(s) which could affect study assessments or may adversely affect the safety and/or success of the study treatment. This includes but is not limited to the following: a. Peripheral neuropathy severe enough to interfere with evaluation of the subject, b. Vascular insufficiency severe enough to interfere with evaluation of the subject, c. Active fibromyalgia, d. Hemiparesis involving either lower extremity, e. Immunocompromised or immunosuppressive disorder or receiving medications to treat immunosuppressive disorders, f. Systemic bleeding disorder(s), g. Current malignancy or treatment within the last 5 years, except for non-melanoma skin cancer, h. Significant psychiatric disorder, i. Active drug and/or alcohol abuse within the past year, j. Uncontrolled diabetes with a Screening Hemoglobin A1C (HbA1c) of >7% k. contraindication to Triamcinolone Hexacetonide (TH) including active tuberculosis, herpes simplex keratitis, acute psychoses and systemic mycoses and paracitoses.
14. Subject is taking medications at the time the subjects signs the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
15. Subject is receiving treatment using electromagnetic stimulation and/or low intensity ultrasound in the Index knee at the time of signing the ICF, within 3 months of signing the ICF or plans to receive treatment any time during the study period.
16. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in Index knee only) corticosteroid within 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the Index knee is allowed.
17. Subject has a pre-treatment contraindication to IA injections or aspiration of the Index knee, including cutaneous infection in the injection site area, active IA infection (as suggested by moderate or marked effusion), knee deformity or condition which, in the opinion of the Investigator could jeopardize the sterility or delivery of the IA injection.
18. Subjects with a history of hypersensitivity to any of the ingredients in the hyaluronan or previous hypersensitivity to the administration of corticosteroids or an inability to tolerate acetaminophen.
19. Subject has any contraindication to the receipt of a corticosteroid.
20. Subject is receiving or in litigation for worker's compensation.
21. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
22. Subject was involved in any other research study involving an investigational product, or a new application of an approved product, within 60 days of signing the ICF.
23. Subject previously treated with Cingal for knee osteoarthritis.

Baseline Exclusion Criteria 25. Subject has a decrease of ≥ 20 mm in the WOMAC pain-sub-score (average of 5 pain scales) from Screening to Baseline in the Index knee on a 100 mm Visual Analog Scale (VAS) scale.

26. Subject has a synovial fluid aspirate volume > 10 mL in the Index knee. 27. Subject has a contraindication to continue with the study treatment injection based on the visual appearance of the synovial fluid aspirate unless the fluid is examined microscopically prior to injection with no clinically significant findings (e.g. bacteria, crystals or blood).

28. Subject has range of motion of less than 100° flexion in either knee.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne MacFie, Study Director — Anika Therapeutics
Locations (26):
- United States (26):
  - Orthopaedic Specialist of North America, PLLC DBA OrthoArizona, Chandler, Arizona
  - Valley Bone and Joint Specialists, Chandler, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Medvin Clinical Research, Covina, California
  - Core Orthopaedic Medical Center (San Dieguito Orthopedic Medical Center), Encinitas, California
  - Infinity Clinical Research, Norco, California
  - Dream Team Clinical Research, Pomona, California
  - Probe Clinical Research Corporation, Riverside, California
  - Artemis Institute for Clinical Research, Riverside, Riverside, California
  - Artemis Institute for Clinical Research, San Marcos, Summerville, California
  - Medvin Clinical Research, Tujunga, California
  - Medvin Clinical Research, Whittier, California
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Shrock Research, Fort Lauderdale, Florida
  - Pines Clinical Research, Inc, Hollywood, Florida
  - Ascension Research, Pinellas Park, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - Anika Therapeutics, Bedford, Massachusetts
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Coastal Carolina Research Center (CCRC), Mt. Pleasant, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Spectrum Medical, Inc., Danville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cingal: Single injection of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH)
- Triamcinolone Hexacetonide (TH): Single injection of a 1 ml dose of Triamcinolone Hexacetonide (TH) containing 20 mg/ml TH
- Placebo: Single injection of a 4 ml unit dose of Placebo containing 0.9% saline
Period: Overall Study
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Started | 99 | 99 | 33
Completed | 99 | 99 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Single injection of a 4 ml dose of Placebo containing 0.9% saline
- Total: Total of all reporting groups
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo | Total
Number analyzed (Participants) | 99 | 99 | 33 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.6) | 58.7 (9.6) | 60.5 (11.3) | 59.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 18 | 141
  Male | 35 | 40 | 15 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 31 | 10 | 66
  White | 70 | 64 | 23 | 157
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Index Knee [Count of Participants; unit: Participants]
  Index Knee - Right | 52 | 45 | 14 | 111
  Index Knee - Left | 47 | 54 | 19 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score
Description: The change from Baseline in knee pain post-treatment as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal arm to the TH arm, the Cingal arm to the Placebo arm, and the TH arm to the Placebo arm. WOMAC Pain is a validated 100 mm visual analog scale (VAS) from 0 mm = No Pain to 100 mm = Highest Pain Level. A negative value for the change from Baseline indicates improvement in the WOMAC Pain Score, i.e. less pain post-treatment. A larger negative value indicates lower pain levels and a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Triamcinolone Hexacetonide (TH): Single injection of a 1 ml unit dose of Triamcinolone Hexacetonide (TH) containing 20 mg/ml TH
- Placebo: Single injection a 4 ml unit dose of Placebo containing 0.9% saline
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -44.3 (21.6) | -37.5 (22.9) | -36.1 (27.8)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.0406, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0795, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.7601, ANOVA

2. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score
Description: The change from Baseline in knee pain post-treatment as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal arm to the TH arm, the Cingal arm to the Placebo arm, and the TH arm to the Placebo arm. WOMAC Pain is a validated 100 mm visual analog scale (VAS) from 0 mm = No Pain to 100 mm = Highest Pain Level. A negative number for the change from Baseline indicates improvement in the WOMAC Pain Score, i.e. less pain post-treatment.
Time Frame: 18 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CINGAL | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -44.5 (21.0) | -40.2 (23.0) | -36.7 (27.0)
Statistical Analysis 1: Comparison: CINGAL vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.1942, ANOVA
Statistical Analysis 2: Comparison: CINGAL vs Placebo; Test type: Superiority; p = 0.0957, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.4526, ANOVA

3. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score
Description: as for outcome 2
Time Frame: 12 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Triamcinolone Hexacetonide (TH): Single injection of a 1 ml unit dose of Triamcinolone Hexacetonide (TH) containing 20 mg/ml of TH
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -44.1 (22.4) | -38.9 (24.5) | -37.4 (25.6)
Statistical Analysis 1: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1309, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1700, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.7609, ANOVA

4. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score
Description: as for outcome 2
Time Frame: 6 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cingal: Single injection a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH)
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -46.0 (23.0) | -40.4 (24.1) | -36.2 (25.1)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.1000, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0423, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.3830, ANOVA

5. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score
Description: as for outcome 2
Time Frame: 3 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -45.1 (21.1) | -37.7 (25.9) | -34.0 (25.5)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.0298, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0217, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.4451, ANOVA

6. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score
Description: as for outcome 2
Time Frame: 1 Week
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -40.9 (22.4) | -35.6 (24.7) | -24.8 (25.4)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.1197, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0008, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.0223, ANOVA

7. Secondary Outcome: The Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index
Description: The post-treatment responder rate is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder to treatment. The criteria for response are (1) improvement in pain or physical function >50% and an absolute change >20 mm; or (2) improvement of >20% with an absolute change >10 mm in at least of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome.
  OMERACT-OARSI responder rates were compared between the Cingal, TH and Placebo arms.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
percentage of participants | 89.9 | 80.8 | 78.8
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.1067, ANOVA

8. Secondary Outcome: Change From Baseline in Knee Pain as Measured by Visual Analog Scale (VAS) Pain Score
Description: Change in knee pain was obtained from participant responses using a 100 mm Visual Analog Scale (VAS) Pain Score at each time point. This VAS scale ranged from 0 mm = No Pain to 100 mm = Highest Pain Level. A negative value for the change in pain indicates less pain post-treatment. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -35.1 (26.0) | -31.9 (25.4) | -27.1 (31.5)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.1715, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0736, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.4098, ANOVA

9. Secondary Outcome: Change From Baseline in Knee Pain as Measured by Numerical Rating Scale (NRS) Pain Score
Description: Change in knee pain was obtained from participant responses using a Numerical Rating Scale (NRS) Pain Score. This NRS Pain Score ranged from 0 = No Pain to 10 = Highest Pain Level. A negative value for the change in Pain Score indicates less pain post-treatment. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -3.5 (2.5) | -3.3 (2.3) | -2.3 (3.1)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.2718, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0182, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.1131, ANOVA

10. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Function Score
Description: The change from Baseline in knee function post-treatment as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Score comparing the Cingal, TH, and Placebo arms. WOMAC Function Score records participant responses regarding the difficulty they have performing daily activities. The WOMAC Function Score is a validated 100 mm visual analog scale (VAS) from 0 mm = No Difficulty to 100 mm = Extreme Difficulty. A negative value for the change from Baseline indicates improvement in WOMAC Function Score. A larger negative value indicates improvement in performing daily activities, and a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -40.8 (23.5) | -37.5 (22.8) | -35.2 (26.5)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.2143, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1628, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.6036, ANOVA

11. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Stiffness Score
Description: The change from Baseline in knee stiffness post-treatment as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Score comparing the Cingal, TH, and Placebo arms. WOMAC Stiffness Score records participant responses regarding the sensation of ease in moving their joint. The WOMAC Stiffness Score is a validated 100 mm visual analog scale (VAS) from 0 mm = No Stiffness to 100 mm = Extreme Stiffness. A negative value for the change from Baseline indicates improvement in WOMAC Stiffness Score. A larger negative value indicates less stiffness, and a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -39.4 (26.0) | -34.6 (25.9) | -32.1 (29.1)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.2220, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1410, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.5418, ANOVA

12. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Total Score
Description: The change from Baseline in overall clinical improvement in the knee post-treatment as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score comparing the Cingal, TH, and Placebo arms. WOMAC Total Score combines the three 0-to-100 point scores from the WOMAC Pain Score, the WOMAC Stiffness Score, and the WOMAC Function Score to calculate a TOTAL Score from 0 = No Symptoms to 100 = Highest Degrees of Pain, Stiffness and Functional Limitation Symptoms.
  A negative value for the change from Baseline in WOMAC Total Score indicates reduction in pain, stiffness, and improved function. A larger negative value indicates a better overall clinical outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -41.4 (22.4) | -37.3 (22.4) | -35.6 (26.2)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.1619, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1683, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.6969, ANOVA

13. Secondary Outcome: Change From Baseline in the Patient Global Assessment (PGA) Score
Description: The change from Baseline in knee pain post-treatment as measured by the Patient Global Assessment (PGA) Score comparing the Cingal, TH, and Placebo arms. PGA Score records participant responses to their assessment of how much their STUDY (treated) knee is bothering them today . The PGA Score is a validated 100 mm visual analog scale (VAS) from 0 mm = No Pain to 100 mm = Extreme Pain.
  A negative value for the change from Baseline indicates improvement in PGA Score. A larger negative value indicates less pain, and a better clinical outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -42.3 (27.3) | -37.6 (25.3) | -34.0 (28.8)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.0701, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.0925, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.6981, ANOVA

14. Secondary Outcome: Change From Baseline in the Evaluator Global Assessment (EGA) Score
Description: The change from Baseline in knee pain post-treatment as measured by the Evaluator Global Assessment (EGA) Score comparing the Cingal, TH, and Placebo arms. EGA Score records the Study Evaluator's assessment of how much the patient's STUDY (treated) knee is bothering them today . The EGA Score is a validated 100 mm visual analog scale (VAS) from 0 mm = No Pain to 100 mm = Extreme Pain.
  A negative value for the change from Baseline indicates improvement in EGA Score. A larger negative value indicates less pain, and a better clinical outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
score on a scale | -40.1 (25.8) | -33.3 (26.0) | -32.6 (24.9)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.0275, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1738, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.8364, ANOVA

15. Secondary Outcome: The Usage of Rescue Medication (Acetaminophen/Paracetamol) at 26 Weeks
Description: The usage of Rescue Medication (RM) as based on the average number of acetominophen/paracetamol pills taken among participants at 26 Weeks post treatment comparing between the Cingal, Triamcinolone Hexacetonide (TH) and Placebo arms.
  A smaller value in average RM indicates that fewer pills were taken by the participants, which may correlate to a better clinical outcome in terms of pain.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
Number analyzed (Participants) | 99 | 99 | 33
Pills | 8.5 (26.1) | 14.2 (31.1) | 19.1 (40.0)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.2227, ANOVA
Statistical Analysis 2: Comparison: Cingal vs Placebo; Test type: Superiority; p = 0.1114, ANOVA
Statistical Analysis 3: Comparison: Triamcinolone Hexacetonide (TH) vs Placebo; Test type: Superiority; p = 0.4635, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of the Baseline Study Visit until Study Completion at 26 Weeks.
Description: The definitions of adverse events and serious adverse events is the same as used in the clinicaltrials.gov definitions.
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Groups:
- Cingal: Single injection of chemically cross-linked sodium hyaluronate supplied as a 4 mL unit dose with a nominal 18 mg of triamcinolone hexacetonide (TH)
- Triamcinolone Hexacetonide (TH): Single injection of TH 20 mg/ml supplied as 1 mL unit dose
- Placebo: Single injection of 0.9% saline supplied as a 4 mL unit dose
Arm/Group | Cingal | Triamcinolone Hexacetonide (TH) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/99 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/99 | 1/99 | 0/33
Other Adverse Events (participants affected / at risk) | 58/99 | 29/99 | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=99) | Triamcinolone Hexacetonide (TH) (N=99) | Placebo (N=33)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Delerium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=99) | Triamcinolone Hexacetonide (TH) (N=99) | Placebo (N=33)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection Site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site joint pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abcess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial food poisoning (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with the conduct of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish Index or the WOMAC® User Guide in any publication, on the Internet or any other public access medium. NICHOLAS BELLAMY, MD, MSc, DSc, MBA, FRACP shall be acknowledged as the source of the Index. Results at the Institution shall not be made before the first multi-site publication by Sponsor. If no multi-site publication within18 months after the Trial completion, PI has right to publish and or present its results (but not the results of any other site) from the Trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT04231318/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT04231318/SAP_001.pdf